CLINICAL TRIAL: NCT04970576
Title: Efficacy of Rivaroxaban in Patients With Left Ventricular Thrombus After Acute Myocardial Infarction: An Open Label Randomized Control Trial
Brief Title: Rivaroxaban in Left Ventricular Thrombus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Jehangir Ali Shah, Associate Professor of Cardiology, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERC-70/2021
Record Dates: First submitted 2021-07-10; First posted 2021-07-21 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Acute Coronary Syndrome; Left Ventricular Thrombus
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Transthoracic echocardiography assessment for the dissolution of LV thrombus will be blinded to the treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Experimental): Patients in the intervention group will receive Rivaroxaban 20 mg once a day (OD) for three months
  Interventions: Drug: Rivaroxaban
- Control group (Active Comparator): Patients in the control group will receive usual warfarin therapy dose adjusted as per the target INR of 2 to 3
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Dose of 20 mg once a day for three months followed by transthoracic echocardiographic assessment for presence/absence of LV thrombus after 4 weeks and 12 weeks
  Arms: Treatment group
Drug: Warfarin — Dose as per the target INR of 2 to 3 with transthoracic echocardiographic assessment for presence/absence of LV thrombus after 4 weeks and 12 weeks
  Arms: Control group

SUMMARY:
The left ventricular (LV) thrombus is an important complication of myocardial infarction (MI) and vitamin K antagonist (VKA) is the current recommended management therapy for these patients. However, lack of regular international normalized ratio (INR) monitoring, drug, and food interaction may leads to increased risk of over or under anticoagulation consequently compromising the effectiveness of the therapy. Hence, due to benefits like predictable dosing and lack of need for regular monitoring, use of non-vitamin K antagonist oral anticoagulants (NOACs) for these patients is increasing among cardiologists. However, clinical data for the justified use of NOACs in LV thrombus (LVT) are lacking and remained a point of debate among the cardiologists. A recently published Randomized Control Trial (RCT) by Abdelnabi M et al. namely the No-LVT trial, had established the safety of Rivaroxaban therapy in patient with post myocardial infarction (MI) LV thrombus along with promising efficacy. However, sample size of the study (n=79; 39 in Rivaroxaban and 40 Warfarin) was not sufficiently high enough to conclude efficacy of Rivaroxaban in these patients. Therefore, this open label RCT is designed with the primary objective to evaluate the efficacy of Rivaroxaban in resolution of post MI LV thrombus as compared to standard warfarin therapy at the interval of 1 month and 3 months to test the hypothesis that Rivaroxaban is safe and non-inferior in preventing thromboembolic and major bleeding events in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of acute coronary syndrome with LV thrombus
* Hemodynamically stable
* Willing to participate

Exclusion Criteria:

* Prior history of cardiomyopathy
* Anticoagulant contraindications
* Prior history of stroke with residual neurological deficit
* Valvular atrial fibrilation
* Pregnancy
* Mentally retarded
* Deranged liver function tests (LFTS)
* Creatinine Clearance <50 ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular (LV) thrombus | After 12 weeks of randomization
  Presence or absence of LV thrombus on transthoracic echocardiographic

SECONDARY OUTCOMES:
Stroke or systemic embolism | Within 12 weeks of randomization
  Confirmed on computerized tomography (CT) scan
Major bleeding | Within 12 weeks of randomization
  As per the International Society on Thrombosis and Haemostasis (ISTH) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jehangir A Shah, FCPS, Principal Investigator — National Institute of Cardiovascular Diseases (NICVD), Karachi, Pakistan
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdelnabi M, Saleh Y, Fareed A, Nossikof A, Wang L, Morsi M, Eshak N, Abdelkarim O, Badran H, Almaghraby A. Comparative Study of Oral Anticoagulation in Left Ventricular Thrombi (No-LVT Trial). J Am Coll Cardiol. 2021 Mar 30;77(12):1590-1592. doi: 10.1016/j.jacc.2021.01.049. No abstract available. PMID 33766266
- [Derived] Shah JA, Hussain J, Ahmed B, Batra MK, Ali G, Naz M, Khan W, Bhatti KI, Karim M, Hakeem A. Rivaroxaban vs Warfarin in Acute Left Ventricular Thrombus Following Myocardial Infarction: RIVAWAR, An Open-Label RCT. JACC Adv. 2025 Aug;4(8):101978. doi: 10.1016/j.jacadv.2025.101978. Epub 2025 Jul 23. PMID 40706143